CLINICAL TRIAL: NCT06523387
Title: Randomized Controlled Trial of an Online Pivotal Response Treatment Training in Autism Spectrum Disorder
Brief Title: Online Pivotal Response Treatment Training in Autism Spectrum Disorder
Acronym: PRT-O
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Grace Gengoux, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-73856
Record Dates: First submitted 2024-07-15; First posted 2024-07-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Pivotal Response Treatment; Parent Training; Online Course
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pivotal Response Treatment Online (PRT-O) Course (Experimental): The PRT-O Online Course (PRT-O) will consist of 10 online lessons completed asynchronously through the Stanford LearnMed Online CANVAS Platform. Parents are expected to view the 10 lessons over the course of a 12-week study period, complete worksheets, and to practice PRT at home.
  Interventions: Behavioral: Pivotal Response Treatment Online (PRT-O) Course
- Delayed Treatment Group (DTG) (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: Pivotal Response Treatment Online (PRT-O) Course — Pivotal Response Treatment - Parent Training
  Arms: Pivotal Response Treatment Online (PRT-O) Course

SUMMARY:
This is a research study that will assess the effects of a Pivotal Response Treatment Online Training Course (PRT-O) for training parents of children with Autism Spectrum Disorder (ASD). The study will specifically investigate whether participants can learn to deliver PRT effectively following participation in the Online training.

ELIGIBILITY:
Inclusion Criteria:

* 2:0 to 5:11 years at the time of consent,
* diagnosed with ASD (based on history, review of available medical records including diagnostic testing, e.g., Autism Diagnostic Observation Schedule) or suspicion of Autism Spectrum Disorder diagnosis, and confirmed with Autism Diagnostic Interview-Revised (ADI-R),
* with significant adaptive communication deficits (i.e., either a Vineland-3 Communication subscale 2 Standard Deviations below average for 2 and 3 year olds and 3 Standard Deviations below for 4 and 5 year olds or a Vineland-3 Expressive V-scale Score 2 Standard Deviations below average for 2 and 3 year olds, or 3 Standard Deviations below for 4 and 5 year old, and at least moderate severity on the Clinical Global Impressions Severity (CGI-S) language subscale),
* an English-speaking parent able to consistently participate in study procedures and conduct treatment in English,
* stable psychotropic medication(s) or biomedical intervention(s) for at least 1 month prior to baseline measurements with no anticipated changes during study participation,
* stable treatment (ABA, Floortime, or other interventions), speech therapy, and school placement for at least 1 month prior to baseline measurements with no expected changes during study participation,
* no more than 60 minutes of 1:1 speech therapy per week

Exclusion Criteria:

* Children who have a primary language other than English
* parent or child diagnosed with severe psychiatric disorder or unstable medical problem
* previous adequate trial of pivotal response treatment resulting in parent meeting Pivotal Response Treatment fidelity of implementation at baseline
* Receiving more than 15 hours of in home 1:1 ABA per week

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on Parent Fidelity of Pivotal Response Treatment Implementation as measured on the Home Video Observation (HVO) | 6 Weeks and 12 Weeks
  Parent Fidelity of Pivotal Response Treatment Implementation will be rated from 10 min HVO by trained coders naïve to treatment assignment and timepoint using established operational definitions from prior PRT studies (e.g., Hardan et al., 2015; Gengoux et al., 2019).
Change from Baseline on Child Functional Verbal Utterances as measures on the Home Video Observation (HVO) | 6 Weeks and 12 Weeks
  Child Functional Verbal Utterances will be rated from 10 min HVO by trained coders naïve to treatment assignment and timepoint using established operational definitions from prior PRT studies (e.g., Hardan et al., 2015; Gengoux et al., 2019).

SECONDARY OUTCOMES:
Change from Baseline on the Clinical Global Impression Scales (CGI) | 6 Weeks and 12 Weeks
Change from Baseline on the Vineland Adaptive Behavior Scales -3 (VABS-3) Communication Domain | 12 Weeks
Change from Baseline on the MacArthur-Bates Communication Scales (CDI) | 12 Weeks

OTHER OUTCOMES:
Change from Baseline on the Stanford Social Dimension Scale (SSDS) | 12 Weeks
Change from Baseline on the Parent Stress Index (PSI) | 12 Weeks
Change from Baseline on the Dimensional Assessment of Repetitive Behavior Scale (DARB) | 12 Weeks
Change from Baseline on the Neurobehavioral Evaluation (NET) Tool | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Grace Gengoux, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No